CLINICAL TRIAL: NCT05450198
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Rising Dose Clinical Trial to Investigate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of MK-6194 in Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Multiple Rising Dose Study of MK-6194 in Participants With Atopic Dermatitis (MK-6194-008)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 6194-008; MK-6194-008 (Other: MSD); 2022-001011-12 (EudraCT Number)
Record Dates: First submitted 2022-07-05; First posted 2022-07-08 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation Panel A (Experimental): Participants are randomized to low dose MK-6194 or placebo, administered every 2 weeks (q2w).
  Interventions: Biological: MK-6194; Biological: Placebo
- Dose Escalation Panel B (Experimental): Participants are randomized to medium dose MK-6194 or placebo administered q2w.
  Interventions: Biological: MK-6194; Biological: Placebo
- Dose Escalation Panel C (Experimental): Participants are randomized to high dose MK-6194 or placebo administered q2w.
  Interventions: Biological: MK-6194; Biological: Placebo
- Expansion Panel D (Experimental): Participants are randomized to medium dose MK-6194 or placebo administered q2w.
  Interventions: Biological: MK-6194; Biological: Placebo
- Expansion Panel E (Experimental): Participants are randomized to a dose less than or equal to high dose MK-6194 or placebo administered q2w.
  Interventions: Biological: MK-6194; Biological: Placebo
- Expansion Dose F (Experimental): Participants are randomized to a dose less than or equal to high dose MK-6194 or placebo q2w.
  Interventions: Biological: MK-6194; Biological: Placebo

INTERVENTIONS:
Biological: MK-6194 — MK-6194 administered subcutaneously (SC)
Biological: Placebo — Placebo comparator to MK-6194 administered SC

SUMMARY:
The primary objective of this study is to characterize the safety and tolerability of MK-6194 following multiple doses among participants with moderate to severe atopic dermatitis who are unresponsive to other therapies.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Clinical diagnosis of atopic dermatitis for at least 6 months prior to the Screening visit.
* Atopic dermatitis is of at least moderate severity.
* History of inadequate response to a stable (≥1 month) regimen of medium to high potency topical corticosteroids or calcineurin inhibitors as treatment for atopic dermatitis within 6 months before the screening visit.
* Body Mass Index (BMI) ≥18 and ≤38 kg/m2 at the screening visit.

Exclusion Criteria:

* Concurrent significant skin disease other than atopic dermatitis (such as psoriasis) or a concurrent clinically significant disease.
* Significant organ dysfunction that is unstable or inadequately treated within 6 months prior to Screening.
* History of cancer (malignancy), with the exceptions: of adequately treated nonmelanomatous skin carcinoma or carcinoma in situ of the cervix or; other malignancies that have been successfully treated with appropriate follow up.
* History of myocardial infarction, congestive heart failure, uncontrolled arrhythmias, cardiac revascularization, stroke, uncontrolled hypertension, or uncontrolled diabetes within 6 months of Screening.
* History of organ or tissue allograft.
* History of symptomatic herpes zoster within 16 weeks of randomization, or any history of disseminated herpes simplex, disseminated herpes zoster, ophthalmic zoster, or central nervous system (CNS) zoster.
* Major surgery within 3 months prior to the screening visit or has a major surgery planned during the study.
* Received a live or attenuated virus vaccine within 4 weeks prior to the Screening visit or intends to receive live or attenuated virus vaccination during the course of the study and for 12 weeks after the last dose of study drug.
* Currently receiving any chronic systemic (oral or intravenous) anti-infective therapy for chronic infection (such as pneumocystis, cytomegalovirus, herpes zoster, or atypical mycobacteria).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (19):
- United States (13):
  - Arkansas Research Trials-Clinical Trials ( Site 0002), North Little Rock, Arkansas
  - Miami Dermatology and Laser Research ( Site 0025), Miami, Florida
  - Global Health Research Center, Inc. ( Site 0005), Miami Lakes, Florida
  - Genesis Clinical Research, LLC ( Site 0004), Tampa, Florida
  - ForCare Clinical Research ( Site 0003), Tampa, Florida
  - Advanced Medical Research, PC. ( Site 0027), Sandy Springs, Georgia
  - AXIS Clinicals ( Site 0029), Dilworth, Minnesota
  - Remington Davis Clinical Research ( Site 0021), Columbus, Ohio
  - Paddington Testing Company ( Site 0010), Philadelphia, Pennsylvania
  - North Texas Center for Clinical Research ( Site 0028), Frisco, Texas
  - Progressive Clinical Research ( Site 0022), San Antonio, Texas
  - Complete Dermatology ( Site 0023), Sugar Land, Texas
  - Premier Clinical Research ( Site 0026), Spokane, Washington
- Anima ( Site 0013), Alken, Limburg, Belgium
- ARENSIA Exploratory Medicine - Sofia ( Site 0018), Sofia, Sofia (stolitsa), Bulgaria
- Innovaderm Research Inc. ( Site 0019), Montreal, Quebec, Canada
- Romania (2):
  - ARENSIA Exploratory Medicine-SC ARENSIA Exploratory Medicine SRL with Monza Medical Center ( Site 00, Bucharest, București
  - ARENSIA Exploratory Medicine-Country Emergency Hospital- Arensia,Cluj-Napoca ( Site 0017), Cluj-Napoca, Cluj
- Hospital Germans Trias i Pujol-CCEE Dermatologia ( Site 0012), Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were enrolled in this study and received MK-6194 or Placebo in Panels A through F. Panels were pre-specified in the protocol to be pooled at dose group level. The exact dose value is proprietary, and directionality is provided.
Groups:
- Placebo: Participants received placebo administered subcutaneously (SC) every 2 weeks (Q2W) in Panels A, B, C, D, E for 7 doses, or every 4 weeks (Q4W) in Panel F for 4 doses.
- MK-6194 Low Dose (Panel A): Participants received low dose of MK-6194 administered SC Q2W for 7 doses.
- MK-6194 High Dose (Panel B-E): Participants received high dose of MK-6194 administered SC Q2W for 7 doses. The dose was the same in Panels B-E and F.
- MK-6194 High Dose (Panel F): Participants received high dose of MK-6194 administered SC Q4W for 4 doses. The dose was the same in Panels B-E and F.
Period: Overall Study
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Started | 18 | 6 | 36 | 12
Completed | 16 | 5 | 32 | 11
Not Completed | 2 | 1 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F) | Total
Number analyzed (Participants) | 18 | 6 | 36 | 12 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (11.0) | 46.5 (11.3) | 42.8 (16.8) | 42.0 (16.5) | 41.6 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 18 | 5 | 30
  Male | 13 | 4 | 18 | 7 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 6 | 1 | 10
  Not Hispanic or Latino | 15 | 6 | 30 | 11 | 62
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 2 | 0 | 3 | 2 | 7
  White | 14 | 6 | 31 | 10 | 61
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Secondary Outcome: Area Under the Curve (AUC) From Days 1-15 (AUC1-15) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the AUC1-15 of MK-6194 in plasma.
Time Frame: Day 1 (Predose and 12 hours postdose), Day 8, and Day 15
Population: The analysis population consisted of all participants who were randomized to MK-6194 and had data available. Samples were excluded if they were at the lower limit of quantification (BLQ) or unevaluable. Samples received thawed were unevaluable. For the Placebo arm, zero participants analyzed indicate data were not generated and no data were available. Panels were pre-specified in the protocol to be pooled at dose group level.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: day*ng/mL
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 2 | 15 | 0
day*ng/mL |  | 32.3 [13.9 to 75.1] | 59.6 [43.8 to 81.1] |

2. Secondary Outcome: AUC From Days 29-43 (AUC29-43) of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the AUC29-43 of MK-6194 in plasma.
Time Frame: Day 29 (Predose and 12 hours postdose), Day 36, and Day 43
Population: The analysis population consisted of all participants who were randomized to MK-6194 and had data available. Samples were excluded if they were at the BLQ or unevaluable. Samples received thawed were unevaluable. For the Placebo arm, zero participants analyzed indicate data were not generated and no data were available. Panels were pre-specified in the protocol to be pooled at dose group level.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: day*ng/mL
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 2 | 20 | 5
day*ng/mL |  | 10.9 [4.13 to 28.7] | 56.7 [41.7 to 77.0] | 86.7 [47.0 to 160]

3. Secondary Outcome: Peak Serum Concentration (Cmax) of MK-6194 (Day 1 to 29)
Description: Blood samples were collected at pre-specified time points to determine the Cmax of MK-6194 in plasma.
Time Frame: Day 1 (Predose and 12 hours postdose), Day 8, Day 15, and Day 29 (Predose and 12 hours postdose)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 4 | 36 | 12
ng/mL |  | 13.2 [6.34 to 27.3] | 21.7 [16.8 to 27.9] | 20.0 [12.9 to 31.1]

4. Secondary Outcome: Minimum Serum Concentration (Ctrough) of MK-6194 (Day 1 to 29)
Description: Blood samples were collected at pre-specified time points to determine the Ctrough of MK-6194 in plasma.
Time Frame: Predose on Days 15 and 29
Population: The analysis population consisted of all participants who were randomized to MK-6194 and had data available. Samples received thawed were unevaluable. For the Placebo arm, zero participants analyzed indicate data were not generated and no data were available. Panels were pre-specified in the protocol to be pooled at dose group level.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 0 | 2 | 0
ng/mL |  |  | 0.210 [0.0141 to 3.13] |

5. Secondary Outcome: Time to Peak Serum Concentration (Tmax) of MK-6194 (Day 1 to 29)
Description: Blood samples were collected at pre-specified time points to determine the Tmax of MK-6194 in plasma.
Time Frame: Day 1 (Predose and 12 hours postdose), Day 8, Day 15, and Day 29 (Predose and 12 hours postdose)
Population: as for outcome 2
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: day
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 4 | 36 | 12
day |  | 0.49 [0.48 to 0.49] | 0.49 [0.48 to 0.51] | 0.49 [0.42 to 0.50]

6. Secondary Outcome: Geometric Mean Accumulation Ratio of AUC of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the geometric mean accumulation ratio of AUC of MK-6194. The accumulation ratio is defined as Day 29-43/ Day 1-15.
Time Frame: Day 1 (Predose and 12 hours postdose), Day 8, Day 15, Day 29 (Predose and 12 hours postdose), Day 36, and Day 43
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 2 | 15 | 0
Ratio |  | 0.35 [0.13 to 0.96] | 0.98 [0.70 to 1.38] |

7. Secondary Outcome: Geometric Mean Accumulation Ratio of Cmax of MK-6194
Description: Blood samples were collected at pre-specified time points to determine the geometric mean accumulation ratio of Cmax of MK-6194. The accumulation ratio is defined as Day 29-43/ Day 1-15.
Time Frame: Day 1 (Predose and 12 hours postdose), Day 8, Day 15, Day 29 (Predose and 12 hours postdose), Day 36, and Day 43
Population: as for outcome 2
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 0 | 4 | 33 | 11
Ratio |  | 0.84 [0.41 to 1.72] | 0.98 [0.79 to 1.20] | 1.35 [0.94 to 1.94]

8. Secondary Outcome: Fold Change From Baseline in Peak Regulatory T Cells (Tregs)
Description: Blood samples were collected to determine the fold change from baseline (FCB) in peak Tregs. The peak Treg FCB was evaluated after the last dose of MK-6194 on Day 85 using natural-log transformed values with a linear model containing fixed effects.
Time Frame: Baseline and Day 85
Population: The analysis population consisted of all participants who were randomized to MK-6194 and had data available. Panels were pre-specified in the protocol to be pooled at dose group level.
Measure: Geometric Least Squares Mean (95% Confidence Interval); unit: Fold change from baseline
Groups:
- MK-6194 Low Dose of (Panel A): Participants received low dose of MK-6194 administered SC Q2W for 7 doses.
Arm/Group | Placebo | MK-6194 Low Dose of (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F)
Number analyzed (Participants) | 16 | 5 | 27 | 11
Fold change from baseline | 1.15 [0.83 to 1.59] | 1.86 [0.95 to 3.66] | 1.69 [1.27 to 2.24] | 1.58 [1.05 to 2.38]

9. Primary Outcome: Number of Participants Who Experience One or More Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 169 days
Population: The analysis population consisted of all participants who received ≥1 dose of study intervention. Panels were pre-specified in the protocol to be pooled at dose group level.
Measure: Count of Participants; unit: Participants
Groups:
- MK-6194 Total: Participants in Panels A through F.
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F) | MK-6194 Total
Number analyzed (Participants) | 18 | 6 | 36 | 12 | 54
Participants | 13 | 6 | 30 | 9 | 45

10. Primary Outcome: Number of Participants Who Discontinue Study Intervention Due to an AE
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study intervention due to an AE is presented.
Time Frame: Up to approximately 85 days
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panel B-E) | MK-6194 High Dose (Panel F) | MK-6194 Total
Number analyzed (Participants) | 18 | 6 | 36 | 12 | 54
Participants | 0 | 1 | 2 | 0 | 3

ADVERSE EVENTS:
Time Frame: Up to approximately 169 days
Description: All-Cause Mortality includes all randomized participants. Serious and Other adverse events (AEs) include all randomized participants who received ≥1 dose of study treatment. Panels were pre-specified in the protocol to be pooled at dose group level.
Groups:
- MK-6194 High Dose (Panels B-E): Participants received high dose of MK-6194 administered SC Q2W for 7 doses. The dose was the same in Panels B-E and F.
Arm/Group | Placebo | MK-6194 Low Dose (Panel A) | MK-6194 High Dose (Panels B-E) | MK-6194 High Dose (Panel F) | MK-6194 Total
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/6 | 0/36 | 0/12 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/6 | 2/36 | 0/12 | 2/54
Other Adverse Events (participants affected / at risk) | 13/18 | 6/6 | 30/36 | 9/12 | 45/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | MK-6194 Low Dose (Panel A) (N=6) | MK-6194 High Dose (Panels B-E) (N=36) | MK-6194 High Dose (Panel F) (N=12) | MK-6194 Total (N=54)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=18) | MK-6194 Low Dose (Panel A) (N=6) | MK-6194 High Dose (Panels B-E) (N=36) | MK-6194 High Dose (Panel F) (N=12) | MK-6194 Total (N=54)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 7 (8) | 3 (5) | 11 (14)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 2 (6) | 1 (1) | 3 (7)
Injection site erythema (General disorders) | 0 (0) | 6 (19) | 25 (110) | 6 (22) | 37 (151)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Injection site induration (General disorders) | 0 (0) | 3 (6) | 8 (16) | 0 (0) | 11 (22)
Injection site oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site pain (General disorders) | 0 (0) | 3 (5) | 6 (7) | 2 (5) | 11 (17)
Injection site pruritus (General disorders) | 0 (0) | 1 (2) | 3 (13) | 0 (0) | 4 (15)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 7 (16) | 3 (5) | 11 (22)
Injection site urticaria (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 3 (4) | 5 (6) | 8 (10)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 5 (6)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypovitaminosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (5) | 1 (1) | 4 (4) | 0 (0) | 5 (5)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embedded device (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Initial insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/98/NCT05450198/Prot_SAP_000.pdf